CLINICAL TRIAL: NCT05790486
Title: Using Rural Community Paramedicine to Engage Lower-Motivated Smokers: Spreading an Effective mHealth-Assisted Intervention to Motivate Cessation
Brief Title: Take A Break - Rural
Acronym: TABR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00087067; 1R01CA268041-01A1 (NIH)
Record Dates: First submitted 2023-03-08; First posted 2023-03-30 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Smoking; Smoking Behaviors; Smoking Cessation
Keywords: smoking rates; public health tobacco control services; smoking cessation service; Rural Health; Implementation Science; Community Paramedicine
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- The Intervention: Take a Break plus Nicotine replacement therapy (NRT) Sampling (Experimental): Motivational text messages, challenge quizzes, goal-setting, coping mini-games, and recognition & rewards. Nicotine lozenges will be given to all participants in both randomized groups.
  Interventions: Behavioral: Take a Break plus Nicotine replacement therapy (NRT) Sampling
- The Comparison: Nicotine replacement therapy (NRT) Sampling without Take a Break (Active Comparator): Nicotine lozenges will be given to all participants in both randomized groups. The goal of the comparison group is to isolate the effect of the Take a Break experience.
  Interventions: Behavioral: The Comparison
- The Enhanced Program: Community Paramedicine Standard Plus Enhanced Implementation Program (Experimental): The Enhanced Program will include strategies described in the Standard Program plus training of local champions.
  Interventions: Other: Community Paramedicine Standard Plus Enhanced Implementation Program
- The Standard Program: Community Paramedicine Standard Implementation Program (Active Comparator): The standard program will include training, resources, and access to the e-refer tool.
  Interventions: Other: Community Paramedicine Standard Implementation Program

INTERVENTIONS:
Behavioral: Take a Break plus Nicotine replacement therapy (NRT) Sampling — Take a Break is an intervention in which smokers are encouraged to engage in smoking abstinence. The main element, the "Break," is a two-week challenge where smokers report days they are smoke-free. The Break is preceded by a 1-week training challenge where Challenge Quizzes (ecological momentary assessments) collect information to guide the smokers during the Break. At baseline, all smokers will be provided NRT lozenges for sampling. At week 1 of the "Marathon", our Tobacco Treatment Specialist will call all smokers, assess their experiences and facilitate an abstinence goal.
  Arms: The Intervention: Take a Break plus Nicotine replacement therapy (NRT) Sampling
Behavioral: The Comparison — The comparison group will receive Nicotine Replacement Therapy sampling and will be balanced in all variables except the Take a Break Intervention.
  Arms: The Comparison: Nicotine replacement therapy (NRT) Sampling without Take a Break
Other: Community Paramedicine Standard Plus Enhanced Implementation Program — Counties randomized to the enhanced program will receive the standard implementation program plus the following enhancements. We will engage and train local implementation champions. The EMS Implementation Champion will go through the Take a Break Intervention but will not receive NRT sampling. The local implementation champions are internal facilitators with additional knowledge and experience related to the electronic referral process. The champions will also be leaders in their county by trying to improve referrals, remind EMS personnel, and distribute feedback on the performance of the county.
  Arms: The Enhanced Program: Community Paramedicine Standard Plus Enhanced Implementation Program
Other: Community Paramedicine Standard Implementation Program — In counties randomized to the standard program, we will engage EMS leaders and train local personnel. The training will be applying the Ask-Advise-Refer model and the use of an eRefer tool in EMS situations and conditions. The EMS will then engage smokers in the field or community to use the Ask-Advise-Refer training to submit electronic referrals with the eRefer tool.
  Arms: The Standard Program: Community Paramedicine Standard Implementation Program

SUMMARY:
The study team proposes a multi-level trial to test 1) novel implementation programs in rural counties designed to increase access to 2) recent advances in tobacco control services for people who are not-yet-ready-to-quit smoking. In this field, most trials have focused only on those already ready-to-quit. Thus, the proposed trial addresses an important knowledge gap critical to advance tobacco control in rural areas.

DETAILED DESCRIPTION:
The study team will conduct a multi-level "hybrid type 2" study (i.e.: implementation and effectiveness outcomes) to test

1) a novel implementation program in rural counties and 2) a mHealth (mobile health)-assisted brief abstinence experience (Take a Break, TAB) for rural adults who smoke and are not-yet-ready to quit. In the network of rural counties, the implementation trial will use a novel, multi-strategy implementation program centered on county employees engaged in 'community paramedicine.' Emergency Medical Services personnel (EMS) are evolving into this more expansive role (e.g.: non-emergent healthcare delivery, monitoring of chronic disease, and preventive medicine). To test the implementation, the study team will randomize rural counties with EMS serving geographically complex and ethnically varied areas (the mountainous region of Appalachia and plains of eastern North Carolina). These counties have some of the highest smoking rates in the U.S. The team will compare a well tested (standard) implementation program versus a novel enhanced program. The standard program uses evidence-based external facilitation - providing training and technical support to EMS services to support the integration of enhanced tobacco control practices (including recommending and referring people who smoke and not-yet-ready-to-quit to the mHealth-assisted population health intervention. The novel enhanced implementation program will include the standard program an EMS Champion program. EMS who currently smoke will be offered participation in TAB themselves. Those who participate, Champions, will then use their TAB experience to support implementation as internal facilitators. They will encourage other EMS to experience TAB, longitudinally encourage use of the tobacco control practices in routine workflow for all EMS, and will be able to use their personal experience with TAB to engage in a richer dialog with patients who smoke. Using these strategies, the team seeks to engage individuals living in harder-to-reach rural areas with less access to clinical services.

Engaging these individuals is possible with brief, low intensity, palatable interventions that target self-efficacy and facilitate skills building to support future abstinence. The TAB intervention addresses the challenge of engaging lower motivated individuals using a novel format, a brief abstinence game, supported using mHealth and building upon 10 years of research. The team recently published the first TAB effectiveness trial in Journal of American Medical Association Internal Medicine. This preliminary data supports the current application and does not include a large number of individuals living in rural areas. In this project, the team will randomize to TAB versus an active comparison designed to isolate the effect of TAB and balance the participant contact across the two groups. In addition to evaluating implementation success and effectiveness outcomes, the team will study pathways to cessation. To inform sustainment and dissemination, the team will collect data on implementation fidelity, county-level adaptations, variations in referrals, and patient-level engagement across the counties, and at the EMS and patient-level. To evaluate budget impact, the team will track the cost of the implementation strategies and the intervention

ELIGIBILITY:
Inclusion Criteria:

* Current Smoker
* at least 18 years old
* speaks English
* Able to receive texts and read text (literate)
* Have a text-enabled phone or receive one from the study team
* Not yet ready to quit smoking

Exclusion Criteria:

* actively quitting smoking
* preparing to quit smoking within 30 days
* prisoners
* FDA- defined NRT contraindications
* unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants engaged | Monthly from initial training to end of referral period year 1 to year 4 longitudinally
  Referral rate of participants by EMS personnel
Follow-up smoking cessation | 6 months
  Point prevalent cessation is measured by the number of participants with a decreased carbon monoxide level as verified by carbon monoxide levels in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Houston, MD, MPH, Principal Investigator — Wake Forest University Health Sciences; Rajani Sadasivam, PhD, Principal Investigator — UMass Chan Medical School
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No